CLINICAL TRIAL: NCT06338670
Title: A Pre-market, Feasibility, Prospective, Open-label, Within Subject Investigation Evaluating the Clinical Performance of the Osia 3 Sound Processor Compared With the Osia 2 Sound Processor in Adult Osia Implant Recipients
Brief Title: Clinical Performance of the Osia 3 Sound Processor Compared With the Osia 2 Sound Processor in Adult Osia Implant Users
Acronym: RECONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5839
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Conductive
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Conductive

STUDY DESIGN:
Intervention Model Description: Within-subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear™ Osia® System (Experimental): Participants will receive the Osia 3 and Osia® 2 sound processors. They will then complete a series of assessments designed to evaluate the clinical performance of these two sound processors. These assessments will take place across four study visits.
  Interventions: Device: Cochlear Osia 3 Sound Processor; Device: Cochlear™ Osia® 2 Sound Processor

INTERVENTIONS:
Device: Cochlear Osia 3 Sound Processor — Osia 3 Sound Processor including sound processor magnets and Osia 3 Aqua +
Device: Cochlear™ Osia® 2 Sound Processor — Osia® 2 Sound Processor and Osia 2 Aqua +

SUMMARY:
This study aims to investigate the clinical performance of the Osia 3 Sound Processor in comparison to the Osia 2 Sound Processor in adults with mixed or conductive hearing loss or single-sided deafness implanted with an Osia implant. Participants will attend four study visits, where they will complete various hearing assessments using the Osia sound processors.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a Cochlear Osia Implant (OSI100 or OSI200)
* Conductive or mixed hearing loss in the implanted ear. Bone conduction threshold 4-frequency pure tone average (PTA4; mean of bone conduction thresholds at 0.5, 1, 2 and 4 kHz) ≤ 55 dB HL.

OR Single-Sided Deafness in the implanted ear. Air Conduction threshold 4-frequency pure tone average (PTA4; mean of air conduction thresholds at 0.5, 1, 2 and 3 kHz) ≤ 20 dB HL in the good ear.

* Aged 18 years or older, at time of consent.
* Minimum experience of 1 month with the Osia 2 Sound Processor.
* Fluent speaker in the language used to assess speech perception performance.
* Willing and able to provide written informed consent.
* For voluntary visit Aqua+ in water only: Be comfortable with going into a swimming pool and putting head under water.

Exclusion Criteria:

* Sensitivity to loud sounds.
* Ongoing infection at or around the sound processor area.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Change (within subject) in speech reception threshold in noise with fixed noise level at 65 dB SPL | During week 48-52
  Speech perception in noise will be measured using the Australian Speech Test in Noise (AuSTIN), which is a test that uses Bamford-Kowal-Bench (BKB)-like target sentences presented in adaptive noise. The AuSTIN corpus comprises 80 lists of 20 sentences each, recorded in female voice. The goal of the adaptive Speech-in-Noise test is to obtain the Speech Reception Threshold in noise.
Change (within subject) in aided thresholds in sound field measured at 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz | During week 48-52
  Aided thresholds in sound field will be measured using warble tones presented from a front speaker positioned at 1 m from the subject following the modified Hughson-Westlake procedure. Frequencies to be tested are 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz.
Change (within subject) in the subjective rating of different aspects of sound when listening to sound clips | During week 48-52
  After listening to different sound clips with Osia 3 and the Osia 2 sound processors, the subjects will rate specific aspects of the sound, e.g., loudness or sound quality, on a Likert scale from 1 to 5 in steps of 1. A rating of 1 is least positive while a rating of 5 is most positive. They will also be asked to explain their sound quality experience in their own words per sound clip.
Change (within subject) in the subjective rating of different aspects of sound during a walk | During week 48-52
  The investigator will hold a conversation with the participant in real-life situations while they wear the Osia 3 sound processor (sound processor only or combined with Osia 3 Aqua+) or Osia 2 sound processor. After the walk, the investigator will ask the participant to rate specific aspects of the sound they experienced on a Likert scale from 1 to 5.
Percentage of participants who preferred Osia 3 over Osia 2 sound processor | During week 48-52
  Participants will be asked which device they prefer after having listened with both devices (Osia 2 and Osia 3) to different sound clips.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Agat, Study Director — Cochlear
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.